CLINICAL TRIAL: NCT03133039
Title: Comparative Experimental and Clinical Study: a New Type of Bioabsorbable Screw and the Titanium Screw in the Hallux Valgus Surgery
Brief Title: A New Type of Bioabsorbable Screw in the Hallux Valgus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Nikke Partio, Resident Surgery (MD), Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R16143
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hallux Valgus; Hallux Rigidus
MeSH Terms: conditions — Hallux Valgus; Hallux Rigidus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioabsorbable screw (Active Comparator)
  Interventions: Procedure: surgery, bioabsorbable screw
- titanium screw (Active Comparator)
  Interventions: Procedure: surgery, bioabsorbable screw

INTERVENTIONS:
Procedure: surgery, bioabsorbable screw — In this study we compare bioabsorbable and titanium screw in the hallux valgus and hallux rigidus surgery

SUMMARY:
The investigators sought to determine whether bioabsorbable cannulated screws could perform as well as titanium cannulated screws in the Lapidus procedure and MTP1-joint arthorodesis in anatomical models and clinical series of the foot.

ELIGIBILITY:
Inclusion Criteria:

* valuntary 18-65-yers-old, patient have hallux valgus or hallux rigidus deformity which need surgery treatment

Exclusion Criteria:

* Over 65 yers-old or less than 18-years-old, diabetes, rheumatism, smoker or lack of co-operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
AOFAS score | 2 years
  score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tampere, Pirkanmaa, Finland